CLINICAL TRIAL: NCT01122771
Title: A Phase III, Open Label, Randomised, Study of Three Short Course Combination Regimens (Ambisome®, Miltefosine, Paromomycin) Compared With AmBisome® Alone for the Treatment of Visceral Leishmaniasis (VL) in Bangladesh
Brief Title: Phase III, Study of Three Short Course Combo (Ambisome®, Miltefosine, Paromomycin) Compared With AmBisome for the Treatment of VL in Bangladesh
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Shaheed Surhawardy Medical College and Hospital (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VLCombo-BD-09
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Visceral Leishmaniasis
Keywords: visceral leishmaniasis; phase III; randomised ccontrolled trial; Bangladesh; Combination treatment; Ambisome; miltefosine; paromomycin
MeSH Terms: conditions — Leishmaniasis, Visceral | interventions — liposomal amphotericin B; miltefosine; Paromomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ambisome (Active Comparator): 15mg Ambisome on days 1,3 and 5
  Interventions: Drug: Liposomal amphotericin B
- Ambisome + Miltefosine (Experimental): Ambisome 5mg + miltefosine 10 days
  Interventions: Drug: liposomal amphotericin B + miltefosine
- Ambisome +paromomycin (Experimental): AmBisome IV infusion (single dose, day 1) + Paromomycin base 11mg/kg/day IM (Gland Pharma, India) for 10 days (days 2-11)
  Interventions: Drug: liposomal amphotericin B + paromomycin
- Miltefosine + paromomycin (Experimental): Oral Miltefosine 1.5-2.5 mg/kg in 1 or 2 doses a day, for 10 days (days 1-10) + Paromomycin base 11mg/kg/day IM for 10 days (days 1-10).
  Interventions: Drug: Miltefosine + Paromomycin

INTERVENTIONS:
Drug: Liposomal amphotericin B — Ambisome i.v. 5mg on days 1, 3 and 5
  Other Names: AmBisome
  Arms: Ambisome
Drug: liposomal amphotericin B + miltefosine — Ambisome 5mg single dose iv Oral Miltefosine 1.5-2.5 mg/kg in 1 or 2 doses a day, for 10 days (days 1-10)
  Other Names: Impavido; AmBisome
  Arms: Ambisome + Miltefosine
Drug: liposomal amphotericin B + paromomycin — Oral Miltefosine 1.5-2.5 mg/kg in 1 or 2 doses a day, for 10 days (days 1-10) + Paromomycin base 11mg/kg/day IM for 10 days (days 1-10).
  Other Names: Impavido
  Arms: Ambisome +paromomycin
Drug: Miltefosine + Paromomycin — Oral Miltefosine 1.5-2.5 mg/kg in 1 or 2 doses a day, for 10 days (days 1-10) + Paromomycin base 11mg/kg/day IM for 10 days (days 1-10).
  Other Names: Impavido
  Arms: Miltefosine + paromomycin

SUMMARY:
This protocol will evaluate the efficacy and safety of various combinations of the three drugs; AmBisome, Paromomycin and Miltefosine at reduced total dosage against the standard treatment with a total dose of 15mg/kg of AmBisome.

DETAILED DESCRIPTION:
Visceral leishmaniasis (VL) is the most severe form of leishmaniasis. The causative parasite in Bangladesh is almost exclusively L. donovani.

• The current treatment options in Bangladesh are not satisfactory as they are either toxic and long, or are of limited use in women of childbearing age due to possible teratogenicity, long treatment duration which leads to non-compliance and possible emergence of resistance or expensive.

In collaboration with Indian Medical Research Council and investigators in India, DNDi initiated a combination trial for treatment of VL in Bihar, India in 2008 including 624 patients from age 5 - 60. The same combinations will be used in the present study. An interim safety review was conducted on the first 120 patients included in the Indian VL Combination study and revealed no safety issues with combination treatment. The enrolment is complete and the final results for 624 patients are expected in Q1 2010.

This is a randomized, controlled, open-label, parallel group study to compare the safety and efficacy of different combination regimens with AmBisome for the treatment of VL in Bangladesh.

This trial is designed in two steps:

Step 1: First 120 patients will be recruited in a hospital setting in a study including parasitology and laboratory assessments at Community Based Medical College, Bangladesh (CBMC,B), primarily for the purpose of reconfirming the safety of combination treatments in Bangladesh. Pending the review and approval of an independent DSMB of the Day 45 data, step 2 will commence.

Step 2: Approximately 554 Patients will then be recruited and treated in Upazilla Health Centre's (UZHC), situated in endemic regions of Bangladesh. We will use rapid diagnostic test (RDT) and the limited laboratory assessments that are available in the centres.

Female patients will be stratified according to marital status, such that unmarried women of child-bearing age will be stratified to receive treatments that do not contain Miltefosine, and married women will be stratified to receive one of the four treatment regimens and must consent to use an approved method of contraception and undergo pregnancy test at the start of the study. Child-bearing age is defined as achieving menarche.

There will be one planned safety review assessing safety and initial cure at Day 45 following completion of Step 1.

ELIGIBILITY:
Inclusion Criteria:

* VL proven by parasitological examination of splenic or bone marrow aspirate. Parasite burden to be graded according to Chulay and Bryceson 1983 and subsequently adopted by WHO. (Step 1 only)
* History of fever, for at least 2 weeks with one or more of the followings criteria: Anaemia (5<Hb<10g/dl), Loss of weight, Splenomegaly
* rk39 positive at baseline assessments
* willing and able to attend follow-up visits
* Male or Female age: 5-60 yrs
* Written informed consent from the patient or from patient's parent or guardian if the patient is under 18 yrs, in addition written assent from patients of 11 - 17 yrs of age. If the patient or parent/guardian are illiterate an impartial witness should be present during the consenting procedure and should also sign.

Exclusion Criteria:

* Married women of child-bearing potential (defined as women who have achieved menarche) who are not using an assured method of contraception or are unwilling to use an assured method of contraception for the duration of treatment and three months after. Assured methods of contraception include i.e. IUCD or depot hormone injection of medroxyprogesterone acetate MPA (DepoProvera®)
* Platelet count less than 40,000/mm3 (Step 1 only)
* Prothrombin time 5 seconds or greater than normal range (Step 1 only)
* Known hepatitis B, C or known HIV positive
* Patients who present with Para Kala-azar Dermal Leishmaniasis
* Signs/symptoms indicative of severe VL (Hb < 5gm/dl, etc)
* Patients with a previous history of VL
* Patients who have received any investigational (unlicensed) drugs within the last 3 months
* Severe malnutrition BMI<15 in adults, weight for height less than 60% in children
* Clinical symptoms of chronic underlying disease such as severe cardiac, renal or hepatic impairment
* Positive HRP2/pLDH Combo test for malaria
* Pregnant woman or breast-feeding mother
* Known alcohol or other drug abuse
* Concomitant chronic drug treatment eg. TB, HIV etc.
* Known hypersensitivity to AmBisome, Paromomycin and other aminoglycosides and/or Miltefosine

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 602 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Definitive cure | 6 month post treatment
  The primary endpoint variable is definitive cure at month 6, and is defined as no significant clinical signs or symptoms of VL at Day 45 including lack of fever [axiliary temperature < 99.5°F] and at least one of the following:
  * improved Hb if the patient was anaemic at baseline (Hb< 8g/dl)
  * spleen regression if the spleen was palpable on admission and absence of clinical signs and symptoms of VL (fever, weight loss, splenomegaly) at any time during 6 months post treatment period.

SECONDARY OUTCOMES:
Initial Cure | Day 45
  Initial Cure is defined as no significant clinical signs or symptoms of VL at Day 45 ie lack of fever [axiliary temp < 99.5°F and at least one of the following:
  * improved Hb if the patient was anaemic at baseline (Hb< 8g/dl)
  * spleen regression if the spleen was palpable on admission
Adverse events | Treatment
  Assess safety during treatment and follow-up in different healthcare settings
  * in hospital setting based on clinical adverse events, laboratory parameters during treatment and 6 months follow-up
  * In UZHC setting based on clinical adverse events, limited laboratory parameters during treatment and 6 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ridwanur Rahman, MD, Principal Investigator — Shaheed Surawardy Medical College
Locations (4):
- Bangladesh (4):
  - Bhaluka UZHC, Bhaluka, Mymensingh
  - Gaffargaon, Gafargaon, Mymensingh
  - Community Based Medical College, Trishal, Mymensingh
  - Trishal UZHC, Trishal, Mymensingh

REFERENCES:
- [Derived] Rahman R, Goyal V, Haque R, Jamil K, Faiz A, Samad R, Ellis S, Balasegaram M, Boer MD, Rijal S, Strub-Wourgaft N, Alves F, Alvar J, Sharma B. Safety and efficacy of short course combination regimens with AmBisome, miltefosine and paromomycin for the treatment of visceral leishmaniasis (VL) in Bangladesh. PLoS Negl Trop Dis. 2017 May 30;11(5):e0005635. doi: 10.1371/journal.pntd.0005635. eCollection 2017 May. PMID 28558062